CLINICAL TRIAL: NCT06089174
Title: Assessment of the Increased Risk of Infection Following an Ultratrail
Acronym: INFultra
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: Jean Monnet University (Other); Hôpital Privé de la Loire- Saint Etienne (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/CHU/23
Record Dates: First submitted 2023-08-11; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Running; Immune Deficiency; Infections
Keywords: Immune deficiency; Ultra-running; Infection
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Infections

STUDY DESIGN:
Intervention Model Description: This study is a descriptive cohort study comparing the occurrence of infection between exposed (runners of an ultra-trail) and unexposed subjects (their companions).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposed (Runners) (Experimental): Ultra-endurance runners taking part in an ultra-trail of 72 km, 109 km or 165 km
  Interventions: Other: Ultra-trail
- Non-exposed (companions) (No Intervention): Runners' companions not running

INTERVENTIONS:
Other: Ultra-trail — Questionnaires sent to runners at various pre-race and post-race times (Day3, Day6, Day10, Day14 and Day21)
  Arms: Exposed (Runners)

SUMMARY:
The increase in the practice of running has encouraged a proliferation of studies evaluating the impact of this sport on health. A number of these studies have looked at the influence of endurance events on the immune system. After prolonged exercise, a systemic inflammatory syndrome sets in, with repercussions for the functioning of the immune system. The number of lymphocytes in the blood is reduced, the function of natural killer (NK) cells is impaired and secretory immunity is impaired. During this period of immunosuppression, often referred to as the 'open window', the host may be more susceptible to micro-organisms that bypass the first line of defence.

The invetigators' hypothesis is therefore that ultratrailers are overexposed to the risk of infection due to immunodepression resulting from practising this sport. In order to support this hypothesis, the investigators would like to look at infectious complications in general and ear-nose and throat episodes (rhinitis, pharyngitis, laryngitis, etc.) in particular, which are the most common infections encountered in primary care, along with urinary tract infections.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Participating in a Grand Raid de la Réunion 2023 race (Mascareignes, Trail de Bourbon, Diagonale des Fous)
* Have a companion living under the same roof during the week preceding the race and the 21 days following the race and who agrees to answer the questionnaires
* Do not object to the research

Exclusion Criteria:

* Do not understand French
* A protected adult (guardianship or curatorship) or under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Increased risk of infection | Day 21
  Comparing the incidence of all infectious symptoms in runners taking part in one of the Grand Raid races (exposed subjects) with the incidence of infectious symptoms in those accompanying them on the race.
  fever, congestion, stuffy nose, sneezing, shortness of breath, vomiting, diarrhea, headache, sore throat, general fatigue, burning and urinary symptoms, other infectious symptoms; associated with major infections (respiratory, skin, gastrointestinal, urinary, other)

SECONDARY OUTCOMES:
Kinetic of infections' appearance | Day 21
  Kinetics of the onset of infectious symptoms within 21 days following one of the Grand Raid de La Réunion races in runners (exposed subjects) and their companions (unexposed subjects). Survival curves over the 3 weeks post-race will be produced.
  An on-line questionnaire will be used to collect infectious data.
Risk factors: running distance | Day 21
  Identify if the distance of the race in which the runner participates is a risk factor associated with the risk of infection in the 21 days following one of the Grand Raid de La Réunion races in runners (exposed subjects).
  An on-line questionnaire will be used to collect data related to the race distance.
Risk factors: training volume | Day 21
  Identify if the runner's training volume is a risk factor associated with the risk of infection in the 21 days following one of the Grand Raid de La Réunion races in runners (exposed subjects).
Risk factors: sex of the runner | Day 21
  Identify if sex of the runner is a risk factor associated with the risk of infection in the 21 days following one of the Grand Raid de La Réunion races in runners (exposed subjects).
Risk factors: age category | Day 21
  Identify if the age of the runner is a risk factor associated with the risk of infection in the 21 days following one of the Grand Raid de La Réunion races in runners (exposed subjects).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BOUSCAREN, MD, Principal Investigator — CHU de la Réunion
Locations (1):
- CHU Réunion, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No